CLINICAL TRIAL: NCT02201459
Title: Randomized Multicenter Phase III Study Comparing the Rate of Molecular Response 4.5 at 12 Months in Newly Diagnosed Philadelphia Positive Chronic Phase Chronic Myelogenous Leukemia Patients Receiving Either Frontline Nilotinib 600 mg Daily or Nilotinib 600 mg Daily Combined to Pegylated Interferon-alfa 2a (Peg-IFN)
Brief Title: Nilotinib ± Peg-IFN for First Line Chronic Phase CML Patients
Acronym: PETALs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013.837
Record Dates: First submitted 2014-06-24; First posted 2014-07-28 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Peg-IFN, nilotinib, MR4.5, CML, chronic phase, first-line
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nilotinib (Active Comparator): Control arm, this compound been licensed in this indication.
  Interventions: Drug: Nilotinib (Tasigna ®), capsules of 150 mg
- Peg-IFN alfa 2a (Pegasys®) and Nilotinib (Experimental): Arm testing the efficacy of a combination of nilotinib and Peg-IFN alfa 2a as frontline therapy for first line chronic phase CML patients.
  Interventions: Drug: Nilotinib (Tasigna ®), capsules of 150 mg; Drug: Nilotinib (Tasigna ®) and Pegylated interferon alfa 2a (Pegasys®)

INTERVENTIONS:
Drug: Nilotinib (Tasigna ®), capsules of 150 mg — Nilotinib 2 capsules of 150 mg orally twice daily at 12 hours difference, fasting (minimum 1 hour before or 2 hours after a meal) for at least 36 months
Drug: Nilotinib (Tasigna ®) and Pegylated interferon alfa 2a (Pegasys®) — * Nilotinib 2 capsules of 150 mg orally twice daily at 12 hours difference, fasting (minimum 1 hour before or 2 hours after a meal) for at least 36 months and
  * Pegylated interferon alfa 2a subcutaneously once a week (auto-injection syringes of 135 and 90 micrograms) at 30 micrograms/week the first month alone (= priming procedure), then at 30 micrograms/2weeks the first month of combination to nilotinib and then at 45 micrograms/week thereafter until month 24 after nilotinib initiation.
  Arms: Peg-IFN alfa 2a (Pegasys®) and Nilotinib

SUMMARY:
This is a phase III trial comparing, for newly diagnosed chronic phase CML patients, nilotinib 600 mg BID as a standard arm and nilotinib 600 mg BID combined to interferon alfa 2 a (pegylated form improving tolerance and maybe enhancing is efficacy) at increased doses for a total of 24 months of combination, in a 1:1 randomized manner. The assessment for the primary efficacy endpoint will be performed at 12 months (since nilotinib initiation) and is the rate patients obtaining MR4.5 will be measured at this time point.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* CP-CML, positive Philadelphia chromosome or positive BCR-ABL (M-bcr transcript), diagnosed less than 3 months prior to study entry
* Age of at least 18 years-old and less than 65 years
* Patient for whom treatment with Nilotinib is expected
* No other CML treatment except for hydroxyurea and/or anagrelide
* No previous TKI treatment.
* No previous treatment with IFN even for other purposes.
* SGOT and SGPT < 2.5 UNL
* Serum creatinine < 2 UNL
* No planned allogeneic stem cell transplantation
* Signed informed consent
* ECOG score 0 to 2

Exclusion Criteria:

* Contra-indication to IFN
* Transcripts other than M-Bcr
* Pregnancy, lactation
* HIV positivity, chronic hepatitis B or C.
* Prior or concurrent malignancy other than CML (exceptions to be mentioned)
* History of arterial occlusive disease or (peripheral, carotids or severe coronary heart disease).
* Permanent elevation of total cholesterol and triglycerides despite treatment
* Severe psychiatric/neurological disease (previous or ongoing)
* Concomitant auto-immune disease
* Other investigational product ongoing
* Ongoing immunosuppressive treatment
* Ongoing treatment at risk for inducing torsades de pointes
* QTcF > 450ms despite correction of predisposing factors (i.e electrolytes…)
* Congenital long QTcF
* Unstabilised thyroid disorder
* No health insurance coverage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Molecular response (MR) 4.5 at 12 months of nilotinib 300 mg twice a day versus a combination of low-dose Peg-Interferon (Peg-IFN) to nilotinib 300 mg twice a day in newly diagnosed CP-CML Chronic Phase Chronic Myelogenous Leukemia patients. | 12 months
  Centralised assessment of the BCR-ABL transcripts at 12 months since nilotinib initiation

SECONDARY OUTCOMES:
Molecular Response 4.5 at 1, 2, 3, 6, 9, 12 months of nilotinib, and duration of MR4.5 during the second year of treatment (18, 24 and 36 months). | 36 months
  Centralised assessment of the BCR-ABL transcripts every month for 3 months and every three months until 12 months and thereafter every 6 months until 36 months assessment.
Major Molecular Response at 1, 2, 3, 6, 9, 12 months of nilotinib, and duration of MMR during the second year of treatment (18, 24 and 36 months). | 36 months
  Centralised assessment of the BCR-ABL transcripts every month for 3 months and every three months until 12 months and thereafter every 6 months until 36 months assessment.
Rate of patients with BCR-ABL/ABL (IS) ≥10% at 3 months. | 3 months after nilotinib initiation
  Centralised assessment of the BCR-ABL transcripts at 3 months.
Rate of CCyR (complete cytogenetic responses: bone marrow Philadelphie positive at 0 % on at least 20 metaphases) at 3, 6, 12 months of nilotinib. | Assessment at 3, 6 and 12 months
  Local bone marrow cytogenetic assessment (on 20 metaphases)
Safety of the nilotinib combined to Peg-IFN or not (hematological and non-hematological adverse events (AE) graded according to the NCI CTC AE v3). | 36 months
  Continuous evaluation of the AEs and SAEs reported during 36 months
Quality of life of patients treated in both arms | 36 months
  EORTC-QLQ C30 and C24 questionnaire at months -1 (Arm B), month 0, 1, 6, 12, 24, 36.
Doses-reductions/interruptions of drugs in both arms. Mean daily doses of nilotinib and Peg-IFN administered. | 24 months for Peg-IFN, and 36 months for both drugs
  Continuous recording of dose intensity along the study for 24-36 months.
Compliance to drugs in each arms | 36 months
  Morisky questionnaire to be fulfilled at 1, 6, 12, 24 and 36 months after nilotinib initiation.
Molecular relapse rate at 6 and 12 months after nilotinib withdrawal in patients obtaining 2-year stable MR4.5. | 36 months
  Local (but standardized) assessment of the BCR-ABL transcripts every months for 3 months.
Event-free survival. | 36 months
  Survival since randomization without any event defined as loss of CHR, loss of PCyR or CCyR, death from any cause, progression towards accelerated phase or blast crisis.
Progression-free survival | 36 months
  Survival without progression towards accelerated of blast phase, death.
Overall survival. | 36 months
  Survival without death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Franck NICOLINI, MD, Principal Investigator — Hopsices Civils de Lyon
Locations (1):
- Franck NICOLINI, Lyon, France

REFERENCES:
- [Background] Abstract We evaluated whether adding pegylated interferon-α2a (Peg-IFNα2a) to nilotinib affected dose intensity, molecular response kinetics, and long-term outcomes in newly diagnosed chronic myeloid leukemia. Delivered nilotinib doses remained comparable between treatment arms up to 72 months, indicating no dose reduction from Peg-IFNα2a-related toxicity. At diagnosis, 8.5 % of 199 patients had additional cytogenetic abnormalities (ACAs). At 3 months, complete and partial cytogenetic response (CCyR/PCyR) rates did not differ between nilotinib alone and the combination (CCyR 72.5 % vs 76 %; PCyR 16.5 % vs 11.5 %). Molecular kinetics showed faster early BCR::ABL1 transcript decline with the combination, but cumulative incidence (CI) curves for major molecular response (MMR) converged by 36 months. Two-year CI of MMR was 80.5 % with nilotinib and 91 % with the combination; five-year CI 93 % vs 97 % (global p = 0.155). The primary endpoint, MR4.5 at 12 months, was reached in 15 % vs 24 % (p = 0.048), but long-term deep molecular response rates (MR4/MR4.5) were ultimately similar at 5 years. In exploratory analyses, female sex (HR 3.06) and higher cumulative Peg-IFNα2a dose in the first 9 months (HR 2.89) predicted early MR4.5, whereas high Sokal or ELTS scores and elevated BCR::ABL1 at month 3 were adverse. ABL1 kinase domain mutations emerged in 10 patients overall (8 nilotinib, 2 combination). Conclusion Peg-IFNα2a with nilotinib accelerated early molecular responses and increased 12-month MR4.5 rates without impairing nilotinib exposure or long-term outcomes. Female sex and Peg-IFNα2a dose intensity correlated with deep early response, supporting potential personalization of combination strategies.